CLINICAL TRIAL: NCT03576118
Title: The Effects of Moderate Versus Deep Neuromuscular Block on Respiratory Mechanics and Biotrauma in Patients With Intraoperative Protective Lung Ventilation for Laparoscopy
Brief Title: Moderate vs Deep Neuromuscular Block on Biotrauma During Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJIRB-MED-OBS-18-115
Record Dates: First submitted 2018-06-14; First posted 2018-07-03 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Pneumoperitoneum
Keywords: biotrauma; laparoscopic surgery; neuromuscular block; sugammadex
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep neuromuscular block (Experimental): Deep neuromuscular relaxation and low pressure pneumoperitoneum
  Interventions: Drug: Deep neuromuscular block
- Moderate neuromuscular block (Active Comparator): Moderate neuromuscular relaxation and standard pressure pneumoperitoneum
  Interventions: Drug: Moderate neuromuscular block

INTERVENTIONS:
Drug: Deep neuromuscular block — Deep neuromuscular block using high dose rocuronium and 8 mmHg pneumoperitoneum
  Other Names: Deep neuromuscular block with rocumeron
  Arms: Deep neuromuscular block
Drug: Moderate neuromuscular block — Moderate neuromuscular block using moderate dose rocuronium and 12-15 mmHg pneumoperitoneum
  Other Names: Moderate neuromuscular block with rocumeron
  Arms: Moderate neuromuscular block

SUMMARY:
The purposes of this study is to investigate the effects of moderate vs. deep neuromuscular block on respiratory mechanics and biotrauma in patients with intraoperative protective lung ventilation for laparoscopy.

DETAILED DESCRIPTION:
Mechanical ventilation results in the disruption of the alveolar-capillary barrier and increased permeability, a hallmark of experimental ventilator-induced lung injury. These mechanical forces also induce an increase in the concentrations of inflammatory cytokines.

The benefits of deep neuromuscular blocks for laparoscopic procedures are controversial and most of the studies undertaken have only sought to improve surgical conditions. Theoretically, deep neuromuscular block permits a lower abdominal insufflation pressure, which leads to better respiratory mechanics and gas exchange. The investigators examined the effects of moderate vs. deep neuromuscular block on respiratory mechanics and biotrauma in patients with intraoperative protective lung ventilation for laparoscopy. The investigators hypothesized that deep neuromuscular block (PTC 1 or 2) and low pressure pneumoperitoneum (8 mmHg) would improve respiratory mechanics and reduce inflammatory processes associated with biotrama during mechanical ventilation compared with moderate neuromuscular block (TOF count 1 or 2 ) and standard pressure pneumoperitoneum (12-15 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II, aged 25 to 80 years, scheduled for laparoscopic surgery with trendelenburg position

Exclusion Criteria:

* cerebrovascular disease
* uncontrolled hypertension, asthma, COPD
* neuromuscular disorder
* patients who have had abdominal surgery
* morbid obesity (body mass index > 35 kg/m2)

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, Principal Investigator — Ajou University Hospital, Suwon, Gyeongki-do, Korea,
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggi-do, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Neuromuscular Block: Moderate neuromuscular relaxation and standard pressure pneumoperitoneum
  Moderate neuromuscular block: Moderate neuromuscular block using moderate dose rocuronium and 12 mmHg pneumoperitoneum
Period: Overall Study
Arm/Group | Deep Neuromuscular Block | Moderate Neuromuscular Block
Started | 37 | 37
Completed | 34 | 33
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Block | Moderate Neuromuscular Block | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (7) | 44 (9) | 44 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 34 | 33 | 67
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of Cytokine
Description: change of IL-6 (pg/ml)
Time Frame: baseline, end of pneumoperitoneum, 24 hr after surgery
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Deep Neuromuscular Block | Moderate Neuromuscular Block
Number analyzed (Participants) | 34 | 33
pg/ml
  IL-6, baseline | 35.9 (16.85) | 12.2 (8.67)
  IL-6, end of pneumoperitoneum | 31.4 (14.85) | 22.9 (9.52)
  IL-6, 24 hr after surgery | 41.53 (16.29) | 32.9 (10.29)

ADVERSE EVENTS:
Time Frame: baseline, end of pneumoperitoneum, 24 hr after surgery
Arm/Group | Deep Neuromuscular Block | Moderate Neuromuscular Block
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03576118/Prot_SAP_000.pdf